CLINICAL TRIAL: NCT00974623
Title: A Prospective Patient Registry for Bone Graft Substitutes in Spinal Fusion: Patient Outcomes and Use in Clinical Practice
Brief Title: Bone Graft Materials Observational Registry
Acronym: APPROACH-001
Status: Terminated | Type: Observational
Why Stopped: Parent sponsor company (Baxter Healthcare) company cut funding
Sponsor: Baxter Healthcare Corporation (Industry)
Collaborators: Apatech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: APPROACH-001
Record Dates: First submitted 2009-09-08; First posted 2009-09-10 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Degenerative Disc Disease; Herniated Disc; Spinal Stenosis; Spondylolithesis; Spinal Deformity; Cervical Myelopathy; Failed Back Surgery Syndrome; Spinal Cord Neoplasms
Keywords: Bone growth substitute; Autograft; Allograft; Spine fusion
MeSH Terms: conditions — Intervertebral Disc Degeneration; Intervertebral Disc Displacement; Spinal Stenosis; Spondylolisthesis; Failed Back Surgery Syndrome; Spinal Cord Neoplasms | interventions — Transplantation, Autologous; Transplantation, Homologous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Spinal Fusion: Patients who undergo a planned spinal fusion procedure requiring approved bone grafting materials (e.g., bone grft substitutes, allograft or autograft).
  Interventions: Device: Bone graft substitute, autograft or allograft

INTERVENTIONS:
Device: Bone graft substitute, autograft or allograft — spine fusion surgery utilizing any commercially available bone graft substitute(s), autograft or allograft
  Other Names: Autograft; Allograft/DBM; Ceramics; Synthetics; BMP; Messenchymal stem cell therapies

SUMMARY:
A multi-center, prospective, observational patient registry to collect information on the clinical outcomes and "real world" use of approved and commercially available bone graft substitutes, autograft and allograft.

ELIGIBILITY:
Inclusion Criteria:

* The patient has failed conservative treatment and is a candidate for spinal fusion surgery.
* The patient is ≥18 years old and of legal age of consent.
* The patient is, in the investigator's opinion, psychosocially, mentally, and physically able to fully comply with this protocol, including the post-operative regimen, required follow-up visits, the filling out of required forms, and have the ability to understand and give written informed consent.
* The patient is skeletally mature (epiphyses closed).
* The patient has signed the IRB approved informed consent.
* The patient is willing and able to participate in post-operative clinical and radiographic follow up evaluations for 2 years.

Exclusion Criteria:

* Patient has systemic infection or infection at the surgical site.
* Patient has a medical condition that would interfere with post-operative assessments and care (i.e., neuromuscular disease, psychiatric disease, paraplegia, quadriplegia, etc.).
* Patient is in poor general health or any concurrent disease process that would place the patient in excessive risk to surgery (i.e., significant circulatory or pulmonary problems, or cardiac disease).
* Patient has a history (present or past) of substance abuse (recreational drugs, prescription drugs or alcohol) that in the investigator's opinion may interfere with protocol assessments and/or with the patient's ability to complete the protocol required follow-up.
* The patient is pregnant/breastfeeding at the time of enrollment, or plans to become pregnant during the course of the study.
* Patient is participating in another investigational study, which could confound results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled in this study will be identified from the surgeon's medical practice and will include patients who failed conservative care and have been identified as requiring spinal fusion surgery.
Sampling Method: Non-Probability Sample
Enrollment: 329 (Actual)
Dates: Start 2009-09; Primary Completion 2013-01 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Evidence of successful radiographic fusion | 6 months, 12 months & 24 months

SECONDARY OUTCOMES:
Maintenance or improvement in neurological status, as compared to baseline scores | 6 months 12 months & 24 months
Improvement of pain/function in comparison to pre-operative QOL scores | 6 months, 12 months & 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Huub Kreuwel, Ph.D, Study Director — Director of Medical Affairs
Locations (14):
- United States (12):
  - UCSF, San Francisco, California
  - St. Joseph's Hospital - Resurgeons Orthopedics, Atlanta, Georgia
  - Carrollton Orthopedics, Carrollton, Georgia
  - Bluegrass Orthopedics & Hand Care Research, Lexington, Kentucky
  - Arthritis & Joint Center - U. Mass. Memorial, Worcester, Massachusetts
  - PRESSD, Southfield, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Montana Neuroscience Institute Foundation, Missoula, Montana
  - Physicians Research Options Spine Center, Las Vegas, Nevada
  - Syracuse Orthopedic Specialists, Syracuse, New York
  - Neurosurgical Associates, Nashville, Tennessee
  - Brain & Spine of Texas, Plano, Texas
- Buda Health Center, Budapest, Hungary
- Isala Klinieken, Groot Wezenland, Zwolle, Netherlands